CLINICAL TRIAL: NCT04904367
Title: The Effectiveness of Deep Tissue Massage on Pain, Trigger Point, Disability, Range of Motion and Quality of Life in Individuals With Myofascial Pain Syndrome
Brief Title: Deep Tissue Massage in the Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer Bingölbali (Other)
Collaborators: Muş Alparslan University (Other)
Responsible Party: Sponsor-Investigator, Ömer Bingölbali, lecturer, Muş Alparslan University
Organization: Muş Alparslan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/306
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Massage Therapy; Myofascial Pain Syndrome
Keywords: Myofascial pain syndrome; Neck disability; Pain; Quality of life
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep tissue massage (Active Comparator): For 4 weeks 20 session, this groups were applied hot pack with 20 minutes of conventional Transcutaneous Electrical Nerve Stimulation(TENS) to back and neck region, followed by 4 minutes of ultrasound at a frequency of 3 Megahertz(MHz) and at a dosage of 1 w / cm2. Also, administered DTM to the back and neck region for 20 min in 12 sessions in addition to the conventional physical therapy.
  Interventions: Procedure: Deep tissue massage; Procedure: Conventional physiotherapy
- Conventional physiotherapy (Experimental): For 4 weeks 20 session, this groups were applied hot pack with 20 minutes of conventional TENS to back and neck region, followed by 4 minutes of ultrasound at a frequency of 3 MHz and at a dosage of 1 w / cm2.
  Interventions: Procedure: Conventional physiotherapy

INTERVENTIONS:
Procedure: Deep tissue massage — The amount of pressure during the massage was adjusted by the physiotherapist with reference to muscle tissue palpation in the patients. During the massage, olecranon, pisiform bone protrusion, metacarpophalangeal and proximal interphalangeal joint faces forearm, wrist and fingers were used during the massage to reach deep tissue. As a massage technique, compression and stretching techniques are used in combination.
  Arms: Deep tissue massage
Procedure: Conventional physiotherapy — For 4 weeks 20 session, this group were applied hot pack with 20 minutes of conventional TENS to back and neck region, followed by 4 minutes of ultrasound at a frequency of 3 MHz and at a dosage of 1 w / cm2.

SUMMARY:
This study aims to examine the effect of deep tissue massage (DTM) on myofascial trigger point (MTrP) number, neck range of motion (ROM), pain, disability and quality of life in patients with Myofacial pain syndrome (MPS).

DETAILED DESCRIPTION:
A total of 88 patients with MPS were screened for eligibility. Of these patients, 80 who met the inclusion criteria were randomly divided into two groups using randomization with computer-generated random numbers as the control group (n=40) and DTM group (n=40).

The patients were evaluated at baseline (Day 0), and the end of treatment (Week 4).

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Have at least one active trigger point
* Have not previously undergone local injectable anesthetic blockage or acupuncture,
* Complaining of pain for the last three months
* Getting a diagnosis of MPS

Exclusion Criteria:

* Patients with infectious skin disease,
* Using analgesic and antidepressant medication,
* A history of major trauma or surgical intervention,
* Mini Mental State Examination (MMSE) score ≤ 24 according

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neck pain on the 10-point Visual Analog Scale(VAS) at 4 week | Baseline and 4 week
  The severity of neck pain was assessed using the visual analog scale (VAS) consists of scores from 0 to 10 in a horizontal line of 10 cm. Patients are asked to mark a place on the scale according to the pain they feel. Increased VAS scores indicate increased pain.
Change from baseline in quality of life on the 36-point Short-Form 36(SF-36) at 4 week | Baseline and 4 week
  Short form-36 (SF-36) was used to determine the quality of life. SF-36, which has a generic scale feature and provides wide angle measurement among the quality of life scales; Ware et al. It was developed and put into use in 1993. The scale includes items including perception of change in health in the last four weeks and perception of change in health in the last week. SF-36 Turkish validity and reliability study has been done. While the increase in the score negatively affects the body pain, physical and emotional role, it positively affects the parameters of physical function, vitality/energy, general health, mental health and social functioning.
Change from baseline in disability on the 20-point at 4 week Neck Pain and Disability Scale (NPDS) at 4 week | Baseline and 4 week
  The Neck Pain and Disability Scale (NPDS) was used for the assessment of disability. This scale was developed by Wheeler et al. NPDS is a 20-item questionnaire developed using VAS as a template. The questions investigate the intensity of pain and its interaction with professional, recreational and functional aspects of life, and the presence and extent of emotional factors related to these. The scoring of each question varies between 0-5. The range of points people can get varies between 0-100. High score values indicate severe disability in patients. NPDS is an index has Turkish reliability and validity, consisting of 20 questions and each question scored between 0 and 5. Increased NPDS scores indicate increased disability.
Change from baseline in range of motion on the universal goniometer at 4 week | Baseline and 4 week
  A universal goniometer was used to evaluate the active neck range of motion (ROM) of the patients. The universal goniometer consists of a pivot point and two arms, fixed and movable. The fixed arm is kept fixed to the immobile part of the extremity or to the floor or body where the measurement is made. The movable arm is the arm that follows and makes the measurement throughout the movement of the measured joint. During our measurement, we chose the pivot point to be the acromion, the earlobe alignment for the movable arm and the fixed arm to be parallel to the ground.
Change from baseline in number of trigger points on the manual palpation at 4 week | Baseline and 4 week
  Manual palpation of the trapezius and levator scapula muscles was performed by a trained physiotherapist in this field to assess the presence of MTrP. Palpation always bilateral was performed with the third and second fingers of each hand with a pressure of no more than 4 kg, which is the conventional approach for detecting tender and trigger points. We considered the pressure of more than 4 kg as whitening of the nail.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer BİNGÖLBALİ, Master, Principal Investigator — Mus Alparslan Universtiy
Locations (1):
- Mus Alparslan University, Muş, Güzeltepe District, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romanowski MW, Spiritovic M, Rutkowski R, Dudek A, Samborski W, Straburzynska-Lupa A. Comparison of Deep Tissue Massage and Therapeutic Massage for Lower Back Pain, Disease Activity, and Functional Capacity of Ankylosing Spondylitis Patients: A Randomized Clinical Pilot Study. Evid Based Complement Alternat Med. 2017;2017:9894128. doi: 10.1155/2017/9894128. Epub 2017 Aug 6. PMID 28845185
- [Background] Kaye AD, Kaye AJ, Swinford J, Baluch A, Bawcom BA, Lambert TJ, Hoover JM. The effect of deep-tissue massage therapy on blood pressure and heart rate. J Altern Complement Med. 2008 Mar;14(2):125-8. doi: 10.1089/acm.2007.0665. PMID 18315516